CLINICAL TRIAL: NCT06713408
Title: Music and Affirmation Recital on Symptom Control, Psychological Resilience and Anxiety Levels
Brief Title: Effects of Music and Affirmation Recital in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-NU-789
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Music
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Music) (Experimental): Audio recordings consisting of pentatonic music and neva makam will be uploaded to the patients' phones by the researcher. Patients will be advised to listen to these music during the period they receive chemotherapy, and they will also be asked to listen to these music in at least 15-20 minute sessions per day and for at least 3 days during the week following chemotherapy.
  Interventions: Other: Experimental (Music)
- Experimental (Affirmation) (Experimental): Patients in this group will be asked to listen to the audio recording with pentatonic music and neva makam in the background, along with the affirmation sentences provided in the appendix. Patients will be advised to listen to these music during the period they receive chemotherapy, and they will also be asked to listen to these music in at least 15-20 minute sessions per day and for at least 3 days during the week following chemotherapy.
  Interventions: Other: Experimental (Affirmation)
- Control (No Intervention): No application will be made to these patients, and standard care practices will be continued.

INTERVENTIONS:
Other: Experimental (Music) — Audio recordings consisting of pentatonic music and neva makam will be uploaded to the patients' phones by the researcher. Patients will be advised to listen to these music during the period they receive chemotherapy, and they will also be asked to listen to these music in at least 15-20 minute sessions per day and for at least 3 days during the week following chemotherapy.
  Arms: Experimental (Music)
Other: Experimental (Affirmation) — Patients in this group will be asked to listen to the audio recording with pentatonic music and neva makam in the background, along with the affirmation sentences provided in the appendix. Patients will be advised to listen to these music during the period they receive chemotherapy, and they will also be asked to listen to these music in at least 15-20 minute sessions per day and for at least 3 days during the week following chemotherapy.
  Arms: Experimental (Affirmation)

SUMMARY:
The aim of this study is to determine the effect of music and affirmation recitals on symptom control, psychological resilience and anxiety levels in women with breast cancer.

DETAILED DESCRIPTION:
Introduction: Music therapy is attracting attention today because it is a person-centered approach that does not require any special skills and/or significant financial investments.

Method: The aim of this study is to determine the effect of music and affirmation recitals on symptom control, psychological resilience and anxiety levels in women with breast cancer. This study will be conducted using a randomized controlled trial design. It is planned to include 75 women in total, 25 patients in the music recital group, 25 patients in the music and affirmation group and 25 patients in the control group. Data in the study will be collected using the Introductory Information Form, Edmonton Symptom Diagnostic Scale, State Anxiety Scale and Psychological Resilience Scale.

Conclusion: It is thought that the findings obtained in this study will contribute to the use of music and affirmation, which are cheap, effective and easily applicable methods, in chemotherapy units as a method to help reduce patients' anxiety. The study is expected to reduce the symptoms of breast cancer patients and reduce their anxiety levels

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with breast cancer
* Those who have received at least 1 course of chemotherapy
* Those over the age of 18
* Those who agree to participate in the study

Exclusion Criteria:

* Those who are not receiving curative chemotherapy
* Those who do not have a phone to listen to music and affirmations
* Those who do not agree to participate in the study
* Those with mental and neuropsychiatric diseases

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Edmonton Symptom Diagnostic Scale | 1 month
  This scale is used to measure cancerous voice, youth, medium units, durable, anxiety, sleepiness, excitement, feeling good and shortness of breath. The measurement of the degree of feeling to be measured from the numbers 0 to 10 on a line on the scale. In the scale, 0 represents no hissing of the symptom, 10 represents very strong hissing. The Turkish validity and publication study of the scale was published by Kurt and Unsar and the Cronbach alpha value works as 0.70.
Beck Anxiety Inventory | 1 month
  Beck Anxiety Inventory: Developed by Beck et al. (1988) to determine the level and frequency of anxiety symptoms experienced by an individual. The scale is a Likert-type self-assessment scale consisting of 21 items and scored between 0-3. The high total score indicates the high level of anxiety experienced by the individual. The score range varies between 0-63. The scale is evaluated as 0-7 points, no anxiety symptoms, 8-15 points, mild anxiety, 16-25 points, moderate anxiety, 26-63 points, severe anxiety symptoms. The validity and reliability study in our country was conducted by Ulusoy et al. (1998) and the Cronbach alpha value of the scale was found to be 0.93.
Brief Resilience Scale | 1 month
  The scale was developed by Smith in 2008, and its Turkish validity and reliability study was conducted by Doğan in 2015. Brief Resilience Scale is a 5-point Likert-type self-report measurement tool consisting of 6 items. The answers are "Not at all appropriate (1), Not appropriate (2), Somewhat appropriate (3), Appropriate (4), Completely appropriate (5)". Items 2, 4, and 6 of the scale are reverse coded. The score obtained from the scale varies between 1 and 30. High scores obtained indicate high psychological resilience. In the validity and reliability study, the Cronbach alpha reliability value of the scale was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

REFERENCES:
- [Derived] Uysal N, Unal Toprak F, Sahingoz Alpargan M. The effect of music and affirmation listening on symptom management, psychological resilience, and anxiety levels in women with breast cancer. Support Care Cancer. 2025 Oct 28;33(11):984. doi: 10.1007/s00520-025-10061-3. PMID 41145719